CLINICAL TRIAL: NCT03105557
Title: Rachitis Device Study
Brief Title: Rickets Device - Feasibility Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Capturin Distribution B.V. (Industry)
Collaborators: Fonds NutsOhra (Other); FrieslandCampina (Industry); Rijnstate Hospital (Other); Scint B.V. (Unknown); Hertog Hendrik BV (Unknown); University of Twente (Other); Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL55778.091.15
Record Dates: First submitted 2017-03-03; First posted 2017-04-10 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Rickets
Keywords: Prematurely born newborns; Urine; Collecting device
MeSH Terms: conditions — Rickets

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Urinary collecting device — Urinary collecting device
  Other Names: Capturin

SUMMARY:
On a daily basis many (prematurely born) newborn are subjected to different urine collecting techniques to study biochemical abnormalities. Neonatology nurses and pediatricians are looking for a better and less invasive manner to collect urine in these vulnerable patients. We hypothesise that the urine collecting device as presented in this protocol is less invasive and has good functional abilities to collect urine in these newborns

Objective of the study:

Clinical feasibility of the urine collection device, indicated by staff and parents.

Study design:

The study will be an open label, clinical feasibility study, of the urine collection device. During a period of 6 months, 30 feasibility tests will be performed.

Study population:

Prematurely born newborns, admitted to the neonatology unit of the department of pediatrics at Rijnstate Hospital Arnhem.

ELIGIBILITY:
Inclusion Criteria:

* Neonates admitted to the neonatology unit of the paediatrics department of Rijnstate Hospital Medical indication for urine testing for Calcium, Phosphate and Creatinine levels Informed consent from parents

Exclusion Criteria:

* No informed consent
* Defective skin in genital region
* Three previous tests in the same subject

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will consist of prematurely born neonates who are admitted to the neonatology unit. And for which the attending physician has an indication to screen for rickets using calcium,phosphate and creatinine level measurement in urine.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2020-01-27 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Questionnaire based clinical feasibility of the urine collection device, indicated by staff and parents | 1 day
  With concern to feasibility we want to know whether this device is able:
  * easy to apply to the neonate
  * to only collect urine
  * to exclude stool admixture
  * easy to use by the nurses
  * comfortable for te neonates

SECONDARY OUTCOMES:
Skin reactions | 1 week
  Number of times skin reactions occurs, reported by the responsible nurse
Skin irritability | 1 week
  Number of times skin irritability occurs, reported by the responsible nurse

CONTACTS AND LOCATIONS:
Locations (1):
- Petra Van Setten, Arnhem, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided